CLINICAL TRIAL: NCT00746590
Title: A Phase 2 Study of the Anti-tumour Activity and Safety of Prolarix™ in Hepatocellular Carcinoma (HCC)
Brief Title: Study of Anti-tumour Effects and Safety of Prolarix™ in Hepatocellular Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated prematurely by sponsor for business reason. One patient was enrolled.
Sponsor: BTG International Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR003-CLN-pro001
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Results first posted 2016-06-09 (Estimated); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; liver cancer; Prolarix; tretazicar; caricotamide; Phase 2; tumor; chemotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Prolarix (tretazicar co-administered with caricotamide)

INTERVENTIONS:
Drug: Prolarix (tretazicar co-administered with caricotamide) — Prolarix (26.6 mg/m2 tretazicar co-administered with 200 mg/m2 caricotamide) administered intravenously every 21 days until disease progression
  Other Names: Prolarix

SUMMARY:
This an open-label study designed to evaluate the anti-tumour activity and safety of Prolarix in subjects with advanced hepatocellular carcinoma.

Prolarix is a chemotherapy comprised of tretazicar as prodrug and caricotamide as co-substrate for the endogenous enzyme, NQO2.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the anti-tumour effects of treatment with Prolarix in subjects with advanced HCC (Child-Pugh A and B only).

All subjects will receive an IV infusion of Prolarix once every 21 days until disease progression is observed.

Subjects will have CT scans for tumour measurements before starting treatment with Prolarix and every 6 weeks until disease progression.

Subjects will undergo evaluation for safety (adverse events, vital signs, clinical laboratory measurements, weight, ECG) every 21 days until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 18 years of age.
* Subject must have a histologic or cytologic diagnosis of HCC and be considered unsuitable for resection or other potentially curative options (eg, liver transplant, curative radiofrequency ablation).
* Subject must have a measurable lesion by RECIST on CT scan in at least one site which has not received radiation or any other local therapy [eg, transcatheter arterial chemoembolisation (TACE), radiofrequency ablation, local injection]. (Note: Subjects who have received local therapies will be allowed to participate, provided that they have a target lesion which has not been subjected to local therapy. Subjects who have received TACE must have a target lesion outside of the vascular territory subjected to chemoembolisation.)
* Subject has an Eastern Cooperative Oncology Group (ECOG) Performance status of 0 or 1.
* Subject has had no other active malignancy within the past three years [other than non melanomatous skin cancer or carcinoma in situ (CIS) of the breast, bladder, or uterine cervix. Subjects with Ta (non-invasive papillary carcinoma) or Tis (sessile carcinoma in situ) bladder cancer are allowed].
* Subject has a minimum life expectancy of at least three months as determined by the investigator.
* Subject has adequate bone marrow function (ie, haemoglobin ≥9 g/dL, granulocytes ≥1500/mm3, platelets ≥75,000/mm3).
* Prothrombin time (PT)-international normalised ratio (INR) ≤2.3 or PT ≤6 seconds above control. (Note: Subjects who are being therapeutically anticoagulated with an agent such as warfarin or heparin will be allowed to participate provided that their INR is between 2.0 and 3.0.
* Subject has adequate renal function (ie, serum creatinine is normal or calculated creatinine clearance is ≥60 mL/min).
* Subject has adequate hepatic function (ie, bilirubin ≤2x upper limit of normal (ULN); AST ALT, and alkaline phosphatase ≤5xULN). (Also see exclusion for Child-Pugh class C below).
* Male subjects and females of childbearing potential must agree to use an adequate method of contraception from the time of initiation of treatment through study participation and for 3 months after release from the study.
* Subject is able to give informed consent.

Exclusion Criteria:

* Any prior or current systemic pharmacotherapy for HCC (cytotoxic, targeted or biologic). (Note: TACE is not considered to be systemic pharmacotherapy for the purpose of this study).
* Subject has an absolute contraindication to receiving CT contrast media. (Note: Subjects with a history of minor contrast reactions may be pre-medicated prior to contrast administration in accordance with local or institutional practice).
* Subject has Child-Pugh Class C hepatic impairment.
* Subject has received an investigational drug within 30 days of enrolment in the study.
* Females of childbearing potential unless using adequate contraception.
* Pregnant or lactating females.
* Major variceal bleeding in the last 30 days.
* Subjects with a known history of human immunodeficiency virus (HIV) infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-09; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claire Daugherty, MS, Study Director — BTG International Inc.
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- Prolarix Treatment Group: Prolarix (tretazicar co-administered with caricotamide): Prolarix (26.6 mg/m2 tretazicar co-administered with 200 mg/m2 caricotamide) administered intravenously every 21 days until disease progression
Period: Overall Study
Arm/Group | Prolarix Treatment Group
Started | 1
Completed | 0
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Prolarix Treatment Group
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Best Tumor Response Rate (Proportion of Subjects With Complete or Partial Response) as Defined by Modified RECIST
Time Frame: every 6 weeks until progression
Population: Study was terminated prematurely after only 1 patient was enrolled. The patient died one month after the initial dose of Prolarix, but his death was unrelated to Prolarix administration.
Measure: Number; unit: Proportion of patients
Groups:
- Prolarix Group: Prolarix (tretazicar co-administered with caricotamide): Prolarix (26.6 mg/m2 tretazicar co-administered with 200 mg/m2 caricotamide) administered intravenously every 21 days until disease progression
Arm/Group | Prolarix Group
Number analyzed (Participants) | 1
Proportion of patients | NA — Study was terminated--the one patient enrolled before termination died after initial dose.

2. Secondary Outcome: Disease Control Rate Defined as the Proportion of Subjects With Either Complete or Partial Response or Stable Disease
Time Frame: Approximately 12 weeks or more after first treatment with Prolarix
Reporting Status: Not Posted

3. Secondary Outcome: Time to Tumour Progression
Time Frame: Every 3 weeks until progression
Reporting Status: Not Posted

4. Secondary Outcome: Post-treatment Changes in the Amount of Contrast-enhancing and Non-contrast-enhancing Tumour
Time Frame: Every 6 weeks until progression
Reporting Status: Not Posted

5. Secondary Outcome: Changes in Alpha Fetoprotein
Time Frame: Baseline, every 3 weeks until progression
Reporting Status: Not Posted

6. Secondary Outcome: Adverse Events
Time Frame: Until progression
Reporting Status: Not Posted

7. Secondary Outcome: Changes in Laboratory Measurements
Time Frame: Baseline and every 3 weeks until progression
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From date of enrollment until the date of death from any cause, assessed every 21 days, up to 1 month.
Description: Study was terminated prematurely - the one patient who enrolled before termination died after their initial dose. This was not related to Prolarix administration.
  Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Prolarix Treatment Group
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prolarix Treatment Group (N=1)
GI toxicity (Gastrointestinal disorders) | 1 (1) — Patient developed GI toxicity resulting in hospitalization considered to be possibly related to study treatment and manifested by dehydration, nausea, anorexia, fatigue, vomiting, diarrhea, and deterioration in performance status (ECOG 3).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No